CLINICAL TRIAL: NCT01587872
Title: Double-balloon Colonoscopy to Increase Cecal Intubation Rate in Technically Difficult Colonoscopies
Brief Title: Double-balloon Colonoscopy to Increase Colonoscopy Completion Rate
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow patient recruitment, not enough patients willing to participate within the prespecified time frame.
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Fujifilm Europa (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SSK_DBC
Record Dates: First submitted 2012-01-12; First posted 2012-04-30 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2012-04

CONDITIONS: Colorectal Cancer; Colorectal Adenomas; Inflammatory Bowel Disease
Keywords: Colonoscopy; Colorectal cancer; Screening colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DBC (Experimental): Double balloon colonoscopy will be attempted in cases where conventional colonoscopy failed due to technical difficulties such as looping or redundant colonic segments.
  Interventions: Procedure: Fujinon EC-450BI5 double-balloon colonoscope

INTERVENTIONS:
Procedure: Fujinon EC-450BI5 double-balloon colonoscope — Colonoscopy with the test instrument

SUMMARY:
The aim of colonoscopy is to visualize the inside of the entire large bowel. Several factors can make the procedure difficult, and sometimes a complete examination is not possible. Complicating factors include poor bowel preparation and technical challenges such as differences in anatomy (long, redundant colonic segments), post-surgical adhesions, strictures and diverticulosis. A special endoscope with two inflatable balloons, originally designed to examine the small bowel, has been used for several years with success in such technically difficult colonoscopies. More recently a modified double-balloon instrument was designed specifically for colonoscopy, but the documentation of the performance of this instrument is limited. The aim of the present study is to investigate the performance of the double-balloon colonoscope in cases where conventional colonoscopy have failed due to technical difficulties.

DETAILED DESCRIPTION:
This is a prospective cohort study to investigate the performance of the test instrument. The test instrument consists of a slim, flexible colonoscope with an overtube and an inflatable balloon on the tip of the colonoscope and the tip of the overtube. Patients are eligible for inclusion if conventional colonoscopy fails due to technical difficulties such as loop formation, long colonic segments or suspected adhesions. Written informed consent is required. The study procedures will be performed immediately after the failed conventional colonoscopy, or on a rescheduled appointment within four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Failed cecal intubation during conventional colonoscopy due to technical difficulties

Exclusion Criteria:

* Failed cecal intubation due to insufficient bowel preparation
* Stenotic colonic lesions
* Patients decline
* Pregnancy
* Persons younger than 18 years
* Persons unable to comprehend the information given

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cecal intubation rate | 2 hours
  The primary outcome measure is a complete or non-complete colonoscopy with the test instrument. Completion is assessed at the end of each procedure.

SECONDARY OUTCOMES:
Detection of additional colonic pathology | 2 hours
  To assess if additional pathology is detected in segments of the colon reached with the test instrument that was not reached with a conventional colonoscope.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bretthauer, PhD, Study Chair — The Cancer Registry of Norway, Oslo University Hospital; Kjetil K Garborg, MD, Principal Investigator — Sorlandet Hospital HF, Kristiansand, Norway
Locations (1):
- Sorlandet Hospital HF, Kristiansand, Norway

REFERENCES:
- [Background] Rex DK, Johnson DA, Anderson JC, Schoenfeld PS, Burke CA, Inadomi JM; American College of Gastroenterology. American College of Gastroenterology guidelines for colorectal cancer screening 2009 [corrected]. Am J Gastroenterol. 2009 Mar;104(3):739-50. doi: 10.1038/ajg.2009.104. Epub 2009 Feb 24. PMID 19240699
- [Background] Neerincx M, Terhaar sive Droste JS, Mulder CJ, Rakers M, Bartelsman JF, Loffeld RJ, Tuynman HA, Brohet RM, van der Hulst RW. Colonic work-up after incomplete colonoscopy: significant new findings during follow-up. Endoscopy. 2010 Sep;42(9):730-5. doi: 10.1055/s-0030-1255523. Epub 2010 Jul 28. PMID 20669092
- [Background] Yamamoto H, Kita H. Enteroscopy. J Gastroenterol. 2005 Jun;40(6):555-62. doi: 10.1007/s00535-005-1645-5. PMID 16007388
- [Background] Moreels TG, Macken EJ, Roth B, Van Outryve MJ, Pelckmans PA. Cecal intubation rate with the double-balloon endoscope after incomplete conventional colonoscopy: a study in 45 patients. J Gastroenterol Hepatol. 2010 Jan;25(1):80-3. doi: 10.1111/j.1440-1746.2009.05942.x. Epub 2009 Aug 3. PMID 19686405
- [Background] Monkemuller K, Knippig C, Rickes S, Fry LC, Schulze A, Malfertheiner P. Usefulness of the double-balloon enteroscope in colonoscopies performed in patients with previously failed colonoscopy. Scand J Gastroenterol. 2007 Feb;42(2):277-8. doi: 10.1080/00365520600802785. No abstract available. PMID 17327949
- [Background] Pasha SF, Harrison ME, Das A, Corrado CM, Arnell KN, Leighton JA. Utility of double-balloon colonoscopy for completion of colon examination after incomplete colonoscopy with conventional colonoscope. Gastrointest Endosc. 2007 May;65(6):848-53. doi: 10.1016/j.gie.2006.08.046. Epub 2007 Feb 26. PMID 17324408
- [Background] Kaltenbach T, Soetikno R, Friedland S. Use of a double balloon enteroscope facilitates caecal intubation after incomplete colonoscopy with a standard colonoscope. Dig Liver Dis. 2006 Dec;38(12):921-5. doi: 10.1016/j.dld.2006.08.003. Epub 2006 Sep 20. PMID 16990055
- [Background] Gay G, Delvaux M. Double-balloon colonoscopy after failed conventional colonoscopy: a pilot series with a new instrument. Endoscopy. 2007 Sep;39(9):788-92. doi: 10.1055/s-2007-966753. PMID 17703387